CLINICAL TRIAL: NCT01890928
Title: Gluconeogenesis Rates and Its Source in Critically Ill Adolescents
Brief Title: Gluconeogenesis Rates and Its Precursors in Pediatric Sepsis
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Texas (Other)
Responsible Party: Principal Investigator, Leticia Castillo, Thomas Fariss Marsh Jr Professor in Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: STU-072010-051
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Sepsis; Hyperglycemia; Critical Illness
Keywords: Gluconeogenesis; Glycogenolysis; Pyruvate cycling; Glucose production rates; Mitochondria; Acylcarnitines
MeSH Terms: conditions — Sepsis; Hyperglycemia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood and urine samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Critically Ill Septic Pediatric Patients: Age 5-12 years; weight ≥ 17kg and Age 13-19 years, males and females
- Healthy Adolescents: Age 13-19 years, males and females

SUMMARY:
Critically ill children have abnormal utilization of nutrients such as glucose, lipids and protein. Often sick children have increased glucose concentrations in blood. However, the origin of the high glucose has not been determined in these populations. There is a close interrelationship between protein and energy metabolism. An increase in the energy supply will not promote nitrogen retention unless the amino acid supply is adequate, and conversely, an increased amino acid supply will be useless if energy is limiting, hence the importance of adequate protein and energy intake. Our study aims to investigate the protein-energy interactions in critically ill septic children and adolescents with the objective to eventually provide the best nutritional support for these patients.

DETAILED DESCRIPTION:
This is an observational study, aimed at exploring:

i) gluconeogenesis rates ii) sources of gluconeogenesis and pyruvate cycling, and iii) protein kinetics in critically ill children and adolescents, and its differences by age group, as well as in comparison to healthy adolescents. The study size will include 45 critically ill septic, pediatric patients (22 children at 5-12 years of age and 23 adolescents' at 13-19 years of age), male and females admitted to the pediatric intensive care unit (PICU) at Children's Medical Center, Dallas. The minimal subject's weight will be 17kg. Additionally, 30 healthy adolescents matched by age, gender, BMI and Tanner stage will be studied at the Clinical Translational Research Center at Zale Lipshy Hospital, to serve as healthy adolescent controls. The number of subjects includes an expected drop out rate of about 20%, in order to obtain 18 patients with complete data in each group. Patients will receive nutritional support as per standard care. This study will yield important knowledge and may lead in the future to changes in the current practice on the management of critically ill pediatric patients in the PICU.

ELIGIBILITY:
Septic Pediatric Patients:

Inclusion Criteria:

1. Children age 5-19 years.
2. Diagnosis of severe sepsis diagnosed as clinical sepsis syndrome (requires two of the following criteria):

   * Source of infection
   * Fever or Hypothermia
   * Leukocytosis or Leucopenia
   * Poor organ perfusion (such as delayed capillary refill or decreased urine output or hypotension)
   * Bacteremic sepsis demonstrated by positive blood culture
3. Indwelling central and/or arterial venous access as per clinical indication.

Exclusion Criteria:

1. Patients with metabolic diseases (i.e.: urea cycle disorders, cystinuria, Insulin dependent diabetes mellitus, etc.).
2. Pregnancy.
3. Primary liver failure.

Healthy Children:

Inclusion Criteria:

1. Age 13-19 years.
2. Evidence of health as assessed by physical exam, and laboratory tests, including: Hematocrit no less than 36% for males and no less than 37% for females, white blood cell count from 5-10,000.
3. Chemistries within normal range, normal urine analysis, and fasting plasma glucose level no less than 60 or greater than 104 mg/dL.
4. Lean Children with BMI of 18-24.
5. Obese Children with BMI of 30 or greater.

Exclusion Criteria:

1. Tobacco use.
2. Pregnancy.
3. Taking any prescription medication that affects amino acid metabolism, i.e., glucocorticoids.
4. History of acute or chronic illness.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Septic pediatric subjects: A total of 45 critically ill children age 5-19 years with diagnosis of sepsis, as defined by the International Sepsis Consensus Conference.
  Healthy subjects: A total of 30 healthy adolescents 13-19 years matched for age, gender, Tanner and BMI to serve as controls. A Dexa scan will be obtained to determine lean body mass.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Gluconeogenesis Rates | 24 hours
  Rates of gluconeogenesis from glycerol, lactate/amino acids in relation to protein synthesis, breakdown and balance, and pyruvate cycling among different age groups (children vs. adolescents) and in comparison with healthy adolescents.

SECONDARY OUTCOMES:
Metabolic Source for Gluconeogenesis | 24 hours during study and overall ICU admission
  Rates of gluconeogenesis from glycerol, lactate/amino acids in relation to severity of the disease, as determined by,
  * PRISM Score III, which is predictor of mortality in pediatric critically ill patients,
  * Degree of inflammation as assessed by plasma C reactive protein,
  * Highest inotrope doses and length of administration,
  * Ventilator-free days, ICU length of stay and length of hospital stay.

OTHER OUTCOMES:
Length of ICU stay | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Castillo, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes